CLINICAL TRIAL: NCT05631548
Title: Identifying Electrophysiological Targets for Transcranial Magnetic Stimulation in Cocaine Use Disorder
Brief Title: Identifying Electrophysiological Targets for Transcranial Magnetic Stimulation in Cocaine Use Disorder (Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Heather E. Webber, PhD, Instructor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC-MS-21-0813 (pilot study)
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cocaine Use Disorder
Keywords: Transcranial Magnetic Stimulation (TMS)

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iTBS to dmPFC, Then Sham iTBS (Experimental)
  Interventions: Device: iTBS to dmPFC; Device: Sham iTBS
- Sham iTBS, Then iTBS to dmPFC (Sham Comparator)
  Interventions: Device: iTBS to dmPFC; Device: Sham iTBS

INTERVENTIONS:
Device: iTBS to dmPFC — TMS will be delivered with a MagVenture Mag Pro R30 with the Cool-B70 A/P coil with active liquid cooling and active/sham sides. Approximately 25% of the nasion-inion distance, or Talairah coordinates X 0 Y+60 Z+60 will be measured.The first session will begin with the acquisition of the resting motor threshold (rMT; lowest stimulus intensity that elicits a visible twitch on 50% of the trials) on the contralateral hand. iTBS (triplet 50 Hz bursts, repeated at 5 Hz, 2 sec on and 8 sec off; 600 pulses per session) will be delivered at 110% of the rMT and will last about 3 minutes. Each participant will receive 2 sessions with a 15-20 minute interval between sessions.
Device: Sham iTBS — Sham TMS will be delivered with the sham side of the MagVenture Cool B70 A/P coil. The software will be pre-programmed by a staff member that will not be involved in data analysis or collection for blinding purposes. The sham stimulation will match the number of pulses and length of time as the active condition and each participant will receive 2 sessions with a 15-20 min interval between sessions.

SUMMARY:
The purpose of this study is to assess the effects of active intermittent theta burst stimulation (iTBS) to dorsomedial prefrontal cortex (dmPFC) on electroencephalogram (EEG) measures of reward sensitivity and cue reactivity and cocaine craving in cocaine users

ELIGIBILITY:
Inclusion Criteria:

* CUD diagnosis

Exclusion Criteria:

* moderate or severe criteria for substances other than cocaine, cannabis, or nicotine
* unstable psychiatric disorder
* medical conditions contraindicated to TMS (e.g., medical implants, history of seizure or seizure disorder, medications lowering the seizure threshold, neurological conditions, moderate-to-severe heart disease)
* pregnancy
* hairstyles incompatible with the EEG net
* head injury with loss of consciousness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Webber, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (2 Sessions)
Arm/Group | iTBS to dmPFC, Then Sham iTBS | Sham iTBS, Then iTBS to dmPFC
Started | 3 | 3
Received Intervention | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — excluded after randomization due to high blood pressure | 0 | 1
Period: Second Interventions (2 Sessions)
Arm/Group | iTBS to dmPFC, Then Sham iTBS | Sham iTBS, Then iTBS to dmPFC
Started | 3 | 2
Received Intervention | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iTBS to dmPFC, Then Sham iTBS | Sham iTBS, Then iTBS to dmPFC | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (9.9) | 37.0 (6.0) | 45.8 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 1 | 0 | 1
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
Years of Education [Mean (Standard Deviation); unit: years] | 12 (0) | 10.5 (1.5) | 11.4 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Amplitude of the Reward Potential (RewP) in Microvolts in Response to Feedback on the Doors Task as Assessed by EEG
Description: The Doors Task will be used to elicit the Reward Potential (RewP) component, representing reward sensitivity. The task is a guessing game, where participants guess which door contains a reward behind it. After selecting a door, the participants are notified if they found the prize by a green arrow pointing up or if they did not find the prize by a red arrow pointing down. The amplitude of the RewP in microvolts in response to feedback is reported.
Time Frame: Baseline (before iTBS session)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
microvolts
  RewP Amplitude with Win | -1.09 (1.95) | 0.61 (1.80)
  RewP Amplitude with Loss | -0.23 (2.15) | 0.12 (1.75)

2. Primary Outcome: Amplitude of the Reward Potential (RewP) in Microvolts in Response to Feedback on the Doors Task as Assessed by EEG
Description: The Doors Task will be used to elicit the Reward Potential (RewP) component, representing reward sensitivity. The task is a guessing game, where participants guess which door contains a reward behind it. After selecting a door, the participants are notified if they found the prize by a green arrow pointing up (win) or if they did not find the prize by a red arrow pointing down (loss). The amplitude of the RewP in microvolts in response to feedback is reported.
Time Frame: Immediately after iTBS session
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
microvolts
  RewP Amplitude with Win | -1.10 (1.54) | 0.21 (1.76)
  RewP Amplitude with Loss | -1.30 (1.05) | 0.02 (1.37)

3. Primary Outcome: Amplitude of the Late Positive Potential (LPP) in Microvolts in Response to Visual Stimuli on the Picture Viewing Task as Assessed by EEG
Description: The Picture Viewing Task will be used to elicit the late positive potential (LPP), reflecting the motivational salience of a stimulus. During this task, participants are asked to view a slideshow of images including pleasant, unpleasant, neutral, and cocaine-related images. The amplitude of the LPP in microvolts in response to visual stimuli is reported.
Time Frame: Baseline (before iTBS session)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
microvolts
  LPP Amplitude with Pleasant Images | 1.10 (1.40) | 0.37 (1.85)
  LPP Amplitude with Unpleasant Images | 1.01 (2.04) | 0.40 (2.55)
  LPP Amplitude with Cocaine Images | .61 (1.49) | 0.46 (1.81)
  LPP Amplitude with Neutral Images | -0.35 (1.51) | -0.95 (2.23)

4. Primary Outcome: Amplitude of the Late Positive Potential (LPP) in Microvolts in Response to Visual Stimuli on the Picture Viewing Task as Assessed by EEG
Description: as for outcome 3
Time Frame: Immediately after iTBS session
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
microvolts
  LPP Amplitude with Pleasant Images | .66 (1.48) | .19 (1.78)
  LPP Amplitude with Unpleasant Images | 1.11 (1.73) | .78 (1.67)
  LPP Amplitude with Cocaine Images | 1.02 (1.31) | .43 (.43)
  LPP Amplitude with Neutral Images | -0.28 (1.21) | -0.0000929 (1.39)

5. Secondary Outcome: Craving as Assessed by the Minnesota Cocaine Craving Scale (MCCS)
Description: The first question (intensity of craving) will be used and is measured from 0(none, not at all) to 100(a great deal), higher number indicating more craving.
Time Frame: Baseline(before iTBS session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
score on a scale | 41 (39.08) | 31.2 (38.55)

6. Secondary Outcome: Craving as Assessed by the Minnesota Cocaine Craving Scale (MCCS)
Description: as for outcome 5
Time Frame: Immediately after iTBS session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
score on a scale | 33.8 (37.81) | 18 (26.39)

7. Secondary Outcome: Pain as Assessed by the Visual Analog Scale (VAS)
Description: This is scored from 0(no pain) to 10 (worst pain), higher score indicating greater pain.
Time Frame: Baseline(before iTBS session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
score on a scale | 0.6 (1.2) | 0.2 (0.4)

8. Secondary Outcome: Pain as Assessed by the Visual Analog Scale (VAS)
Description: This is scored from 0(no pain) to 10 (worst pain), higher score indicating greater pain.
Time Frame: Immediately after iTBS session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
score on a scale | 2 (3.52) | 1.6 (1.74)

9. Secondary Outcome: Cognitive Function as Assessed by the Montreal Cognitive Assessment (MoCA)
Description: Total score on the Montreal Cognitive Assessment (MoCA) range from 0 to 30, with a higher score indicating a better outcome.
Time Frame: Baseline(before iTBS session)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
score on a scale | 23 (4.05) | 22.8 (4.96)

10. Secondary Outcome: Cognitive Function as Assessed by the The Montreal Cognitive Assessment (MoCA)
Description: as for outcome 9
Time Frame: Immediately after iTBS session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iTBS to dmPFC | Sham iTBS
Number analyzed (Participants) | 5 | 5
score on a scale | 22.4 (3.01) | 25 (2.76)

ADVERSE EVENTS:
Time Frame: from baseline until study completion (i.e., 2 weeks)
Arm/Group | iTBS to dmPFC | Sham iTBS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | iTBS to dmPFC (N=5) | Sham iTBS (N=5)
Scalp Discomfort (General disorders) | 2 | 1
Neck Pain (General disorders) | 1 | 0
Headache (General disorders) | 2 | 0
Muscle Spasm (General disorders) | 1 | 0
Light-Headed (General disorders) | 1 | 1
Tingling (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT05631548/Prot_SAP_000.pdf